CLINICAL TRIAL: NCT05217433
Title: A Randomized, Double-blind, Placebo Controlled Study to Investigate the Efficacy of Oleuropein on Skeletal Muscle Energy Metabolism and Fatigue in Humans
Brief Title: Oleuropein and Muscle Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20.22.NRC
Record Dates: First submitted 2021-11-25; First posted 2022-02-01 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Muscular Fatigue
Keywords: Skeletal muscle energy and fatigue
MeSH Terms: conditions — Fatigue | interventions — olive leaf extract

STUDY DESIGN:
Intervention Model Description: This is a single-centre, double-blind, placebo controlled, randomised 2-arms parallel group study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a single-centre, double-blind, placebo controlled, randomised 2-arms parallel group study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational product (Experimental): The investigational product is a capsule containing 100mg of the active ingredient oleuropein and will be provided once daily in the form of a 250mg olive leaf extract (i.e. 100mg of oleuropein per day) product for the duration of the intervention period (36 days).
  Interventions: Other: Olive leaf extract
- Control arm (Placebo Comparator): The control will be a placebo capsule containing 336 mg of cellulose microcrystalline, matching the investigational product appearance.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Olive leaf extract — The investigational product is a capsule containing 100mg of the active ingredient oleuropein and will be provided once daily in the form of a 250mg olive leaf extract (i.e. 100mg of oleuropein per day) product for the duration of the intervention period (36 days).
  Arms: Investigational product
Other: Placebo — The control will be a placebo capsule containing 336 mg of cellulose microcrystalline, matching the investigational product appearance.
  Arms: Control arm

SUMMARY:
Preclinical studies performed at Nestlé Research (NR) identified oleuropein as a novel activator of mitochondrial calcium import. This potentiated mitochondrial calcium uptake resulted in decreased phosphorylation of the enzyme pyruvate dehydrogenase (PDH), which is linked to its activation as a rate limiting enzyme for mitochondrial oxidation, as well as increasing mitochondrial oxygen consumption, resulting ultimately in decreases in muscle fatigue. In addition, NR demonstrated that during aging, mitochondrial calcium and oxygen consumption rates are decreased in isolated skeletal muscle fibers. The next step in the evidence development is to demonstrate efficacy of oleuropein for improved muscle energy and decreased physical fatigue in a healthy aging population.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. 50 to 70 years old
3. BMI 18.5-29.9 kg/m2
4. Healthy as per medical history and investigator's/ physician's judgement
5. Having given informed consent

Exclusion Criteria:

1. Allergy/intolerance to the study product
2. >5% body mass change in the previous 3 months
3. HbA1c ≥ 6.5%
4. Blood pressure >140/90 mmHg
5. Participating in a structured (progressive) exercise program
6. Smoking
7. Diagnosed acute or chronic medical conditions that, in the opinion of the investigator, could impact study outcomes
8. Diagnosed musculoskeletal disorders
9. Chronic use of gastric acid suppressing medication
10. Unauthorized concomitant medications such as calcium antagonists (e.g. valproate), oral corticosteroids, anything that will prevent subjects from safely completing the study according to the investigator or medications / drugs known interfering with the expected mechanism of action of IP or to affect the outcome parameters
11. Alcohol (intake higher than 3 servings per day. One serving is 0.4 dl of alcohol, 1 dl of wine, or 3 dl of beer) or drug abuse
12. Overly imbalanced or restrictive diet (e.g. hyperproteic, vegan, ketogenic, etc.)
13. Subjects not willing and/or not able to comply with scheduled visits and the requirements of the study protocol
14. Any implants that would be a contra-indication for performing an MRI scan.
15. Participation in another study at the same time
16. Blood donation in the past 2 months

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 1. Male
  2. 50 to 70 years old
  3. BMI 18.5-29.9 kg/m2
  4. Healthy as per medical history and investigator's/ physician's judgement
  5. Having given informed consent
Enrollment: 40 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Exploratory outcomes - Evaluate the changes in Pyruvate dehydrogenase activation between oleuropein and placebo groups following 1 single dose | Chronic effect after 36 days of intake
  measured by western blotting
Exploratory outcomes - Evaluate the changes in Pyruvate dehydrogenase activation between oleuropein and placebo groups following 1 single dose | Acute effect after first product intake + chronic effect after 36 days of intake
  measured by biochemical assay analysis
Exploratory outcomes - to evaluate the changes Mitocondrial respiration between oleuropein and placebo groups following 1 single dose | Acute effect after first product intake + chronic effect after 36 days of intake
  measured the rates of oxygen consumption (respiration or JO2) using Oroboros Oxygraph 2K systems with physiological ADP concentrations using permeabilized muscle fibres.
Exploratory outcomes- to evaluate the changes of fatigue between oleuropein and placebo groups following 1 single dose | After 4 weeks of supplementation
  measured using Biodex dynamometer
Exploratory outcomes - to evaluate the changes of fatigue between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  measured using Biodex dynamometer
Exploratory outcomes - to evaluate the changes of Pyruvate dehydrogenase activation between oleuropein and placebo groups | Chronic effect (after 36 days of supplementation)
  measured by western blotting
Exploratory outcomes - to evaluate the changes of Pyruvate dehydrogenase activation between oleuropein and placebo groups | Chronic effect (after 36 days of supplementation)
  measured by biochemical assay analysis
Exploratory outcomes - To evaluate the changes of Mitochondrial respiration between oleuropein and placebo groups | Chronic effect (after 36 days of supplementation)
  measured the rates of oxygen consumption (respiration or JO2) using Oroboros Oxygraph 2K systems with physiological ADP concentrations using permeabilized muscle fibres.

SECONDARY OUTCOMES:
Exploratory outcomes - to evaluate the changes of whole body respiratory exchange ratio (RER) between oleuropein and placebo groups following 1 single dose | Acute effect after first product intake+ chronic effect after 36 days of intake
  measured the oxygen and carbon dioxide volume using indirect calorimetry with ventilated hood
Exploratory outcomes - to evaluate the changes of oleuropein metabolites between oleuropein and placebo groups following 1 single dose | Acute effect after first product intake + chronic effect after 36 days of intake
  measured by the analyze of oleuropein metabolites in blood
Exploratory outcomes - to evaluate the changes of glucose concentration between oleuropein and placebo groups following 1 single dose | Acute effect after first product intake + chronic effect after 36 days of intake
  measured by the analyze glucose in blood
Exploratory outcomes - to evaluate the changes Blood glucose, insulin, free fatty acid concentrations -between oleuropein and placebo groups following 1 single dose | Acute effect after first product intake + chronic effect after 36 days of intake
  measured by the analyze of Insulin in blood
Exploratory outcomes - to evaluate the changes of free fatty acid concentration between oleuropein and placebo groups following 1 single dose | Acute effect after first product intake + chronic effect after 36 days of intake
  measured by the analyze of free fatty acid concentration (FFA, TG) in blood
Exploratory outcomes - to evaluate the changes of blood pressure between oleuropein and placebo groups following 1 single dose | Acute effect after first product intake + chronic effect after 36 days of intake
  measured using automated inflatable cuff
Exploratory outcomes - to evaluate the changes of anti-inflammatory markers between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  measured by the analyze of anti-inflammatory markers in blood
Exploratory outcomes - to evaluate the changes of Antioxidant markers between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  measured by the analyze of antioxidant markers in blood
Exploratory outcomes - to evaluate the changes in glucose concentration between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  measured by the analyze glucose in blood
Exploratory outcomes - to evaluate the changes of insulin concentration between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  measured by the analyze of insulin in blood
Exploratory outcomes - to evaluate the changes of free fatty acid concentration between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  measured by the analyze of free fatty acid concentration (FFA, TG) in blood
Exploratory outcomes - to evaluate the changes in Mood state and quality of life between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  measured with the World Health Organisation quality of life questionnaire (WHOQOL-BREF) (rating 0 for 'not at all' and 5 for 'an extreme amount')
Exploratory outcomes - to evaluate the changes in Mood state and quality of life between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  measured with the Profile of Mood States - short-form (POMS-SF) - scale (rating 0 for 'not at all' and 4 for 'extremely')
Exploratory outcomes - to evaluate the changes in Mood state and quality of life between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  measured with the Quality of Life (QoL) questionnaires
Exploratory outcomes - to evaluate the changes in the fatigue perception and mood state pre/post Biodex measurement between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  measured with the current mood questionnaire (rating 0 for 'not at all' - 4 for 'extremely')
Exploratory outcomes - to evaluate the changes in the fatigue perception and mood state pre/post Biodex measurement between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  RPE visual analog scale Questionnaire - BORG scale (6 for 'no exertion - 20 for 'maximal exertion'
Exploratory outcomes to evaluate the changes in body composition between oleuropein and placebo groups | Chronic effect (after 29 days of supplementation)
  measure the whole body muscle and fat content using Magnetic resonance imaging (MRI)
Exploratory outcomes - Whole body respiratory exchange ratio - To evaluate the changes of Whole body respiratory exchange ratio (RER) between oleuropein and placebo groups | Chronic effect (after 36 days of supplementation)
  measure the oxygen and dioxygen volume using Indirect calorimetry with ventilation hood
Exploratory outcomes - To evaluate the changes of oleuropein metabolites between oleuropein and placebo groups | Chronic effect (after 36 days of supplementation)
  measure by analyzing Oleuropein metabolites in blood
Exploratory outcomes - to evaluate the changes of molecular signalling, and protein and mRNA levels of regulators of muscle metabolism between oleuropein and placebo groups | Chronic effect (after 36 days of supplementation)
  measured by analyzing RNAseq and MS-based proteomics
Exploratory outcomes - to evaluate the changes of molecular signalling, and protein and mRNA levels of regulators oleuropein and placebo groups | Chronic effect (after 36 days of supplementation)
  measured using Western Blot
Exploratory outcomes - to evaluate the changes of molecular signalling, and protein and mRNA levels of regulators oleuropein and placebo groups | Chronic effect (after 36 days of supplementation)
  measured by analyzing polymerase chain reaction
Exploratory outcomes - to evaluate the changes in Strength between oleuropein and placebo groups | After 4 weeks of supplementation
  measured using biodex dynanometer
Exploratory outcomes to evaluate the changes of strenght between oleuropein | Chronic effect (after 29 days of supplementation)
  measured using biodex dynanometer

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Centre +, Maastricht, Netherlands

REFERENCES:
- [Derived] Pinckaers PJ, Petrick HL, Horstman AM, Moreno-Asso A, De Marchi U, Hendriks FK, Kuin LM, Fuchs CJ, Grathwohl D, Verdijk LB, Zorenc AH, Senden JM, Migliavacca E, Metairon S, Poquet L, Morin-Rivron D, Karagounis LG, Holloway GP, Feige JN, van Loon LJ. Oleuropein Supplementation Increases Resting Skeletal Muscle Fractional Pyruvate Dehydrogenase Activity but Does Not Influence Whole-Body Metabolism: A Randomized, Double-Blind, and Placebo-Controlled Trial in Healthy, Older Males. J Nutr. 2025 May;155(5):1373-1386. doi: 10.1016/j.tjnut.2025.02.015. Epub 2025 Feb 22. PMID 39993475